CLINICAL TRIAL: NCT03953963
Title: Evaluation of the Removal of Excess Intra-Abdominal Fat in Subjects With Type 2 Diabetes and Obesity, Using the HydraSolve T2D™ System, on Glucose Control, Insulin Resistance and Body Weight
Brief Title: Evaluation of Intra-Abdominal Fat Extraction Using HydraSolve T2D™ in Obese Subjects With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medality Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-00001
Record Dates: First submitted 2019-05-12; First posted 2019-05-17 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Mesenteric Visceral Fat; Insulin Resistance; Diabetes; Type 2 diabetes; Diabetes Mellitus; Noninsulin-Dependent Diabetes Mellitus; Glucose Metabolism Disorder; Obesity; Diabesity; HydraSolve T2D
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus; Glucose Metabolism Disorders; Obesity; Diabesity

STUDY DESIGN:
Intervention Model Description: Patients will be experimental subjects, they will serve as their own controls by comparing their pre-op status to their post-op status in the parameters of investigation which include insulin status assessment (resistance versus sensitivity, as determined by hyperinsulinemic euglycemic clamp), measurements of glycemic control of T2D, and body weight measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intra-Abdominal Mesenteric Fat Extraction Group (Experimental): All enrolled patients will undergo the combined minimally invasive laparoscopic and mini-laparotomy procedure to selectively extract excess intra-abdominal fat from the mesentery.
  Interventions: Device: HydraSolve T2D™

INTERVENTIONS:
Device: HydraSolve T2D™ — The HydraSolve T2D™ System will be used to perform the combined minimally invasive laparoscopic and mini-laparotomy procedure to selectively extract excess intra-abdominal fat from the mesentery. All patients will receive standard nutritional counseling and their medications will be adjusted to achieve target levels of blood glucose control.

SUMMARY:
This study will investigate the safety and efficacy of the investigational use of the HydraSolve T2D™ System in improving blood glucose control and insulin resistance in patients with obesity (Class 1, BMI 30-39.9 kg/m2) and type 2 diabetes who have not achieved targeted levels of blood glucose control using oral diabetes medications. The previously FDA-cleared (for liposuction and fat transfer) HydraSolve T2D™ System will be used to perform a novel, minimally invasive laparoscopic and mini-laparotomy procedure to selectively remove excess intra-abdominal fat from the mesentery (Mesenteric Visceral Lipectomy (MVL)), while not affecting surrounding tissues. The study will include several weeks of screening for eligibility before the intervention, and 12-months of follow-up post-surgery.

DETAILED DESCRIPTION:
This study will evaluate the investigational use of the HydraSolve T2D™ System (previously FDA-cleared for liposuction and fat transfer) to perform a novel, minimally invasive laparoscopic and mini-laparotomy procedure to selectively remove intra-abdominal fat from the mesentery and to assess the resulting changes in blood glucose control, insulin sensitivity and body weight. Excess intra-abdominal mesenteric fat has been directly linked to insulin resistance, an important precursor of type 2 diabetes. Up to 30 study candidates will undergo screening and eligibility testing over a 5-week period from which 12 will be enrolled to undergo the procedure. During the 12-month period post-procedure, the patients will be periodically monitored for improvements in blood glucose control (HbA1c, oral glucose tolerance test (OGTT), fasting blood glucose (FBG) and continuous glucose monitoring (CGM)), insulin resistance (hyperinsulinemic euglycemic glucose clamp), body weight, changes in fat deposits (Magnetic Resonance Imaging (MRI) and Magnetic Resonance Spectroscopy (MRS) and Dual-Energy X-ray Absorptiometry (DEXA)) and overall metabolic health (including indirect calorimetry and various biomarkers). This prospective, single-arm study uses pre-operative patient data as the control. Safety assessments and monitoring for adverse events will be performed, throughout.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willingness to provide written informed consent.

  2. Willingness and availability to comply with study requirements for the duration of the study, including specific inquiry that the potential subject does not have an impending move or travel planned and can attend the patient visits without undue hardship.

  3. Male or female between 22 - 75 years of age. (Caveat: premenopausal women are excluded)

  4. In good general health except for being diagnosed as having T2D,and in good enough general health to undergo a conversion from a mini-laparotomy to an open laparotomy incision if that conversion becomes necessary during the operative procedure; the subject has no major system disease other than T2D as determined by physical examination, medical history, screening laboratory tests, and EKG.

  5. BMI 30 to 39.9 kg/m2.

  6. Stable body weight during the 6 month time period preceding the anticipated surgery date. (Stable is defined as: the usual baseline body weight of the subject +/- < 5% change.)

  7. Diagnosis of T2D 10 years or less in duration.

  8. Subject has poorly controlled T2D and is on a current regimen of at least two oral hypoglycemic agents, the first medication dosed at the maximum dose, and the second dosed at the minimum or higher labelled dose. Subject's treatment regime does not include insulin treatment.

  9. HbA1c: 8.0 % - 10.0 %, taken within 30 days pre-op.

  10. Subjects receiving exogenous thyroid hormone, a euthyroid status for at least 3 months prior to enrollment needs to be documented.

  11. Subject agrees to not take any medications that can influence glycemic control unless directed to do so specifically by their physician.

  12. Subject agrees to report all medications they are taking on all case report forms.

  13. Subject agrees to not take any herbal or dietary supplements during the study period.

  14. Subject agrees to not donate blood during the study period.

  15. Subject resides in the San Antonio, TX geographic area.

  16. Subject is able to have MRI examinations.

Exclusion Criteria:

* 1. Premenopausal females.

  2. Tobacco use.

  3. Current drug or ETOH abuse.

  4. Uncontrolled psychiatric illness.

  5. Abnormal T4 and TSH found in screening blood test.

  6. Subjects who have contraindications to major abdominal surgery are excluded.

  7. Serum albumin <35 g/L

  8. Body weight loss >5% during the 6 month time period preceding the anticipated surgery date.

  9. Presence of a remote body site infection. (Examples: dental urinary, skin soft tissue)

  10. History of cholecystitis, hepatitis or NASH.

  11. History of ulcerative colitis, Crohn's disease, or diverticulitis.

  12. History of respiratory conditions that are not controllable without the use of chronic or intermittent steroid use; such as poorly controlled asthma or COPD.

  13. Chemistry, liver enzyme and function, and hematology levels that are outside of the normal range. (Fasting glucose may be elevated but subject will be excluded if it is ≥ 250 mg/dl.)

  14. LDL ≥ 180 mg/dl.

  15. Triglycerides ≥ 400 mg/dl.

  16. A diagnosis of Cushing's disease. (If a potential subject does not have a diagnosis of Cushing's disease, and the examining endocrinologist detects concerning signs or symptoms that lead him/her to suspect that the potential subject may have Cushing's disease (based on the subject's history, review of systems and physical exam) then that potential subject will be excluded from the study and referred back to his/her primary care physician for further evaluation.)

  17. Anemia, hemoglobinopathy or any conditions that increase red blood cell turnover.

  18. Recent history of receiving a blood transfusion.

  19. Recent history of donating blood.

  20. Clinically significant major organ disease as determined by medical history, physical exam, screening blood tests, urinalysis, and EKG.

  21. History of prior abdominal/pelvic surgery, or prior OB/GYN surgery.

  22. Uncontrolled comorbidity. (Example: uncontrolled hypertension.)

  23. Large umbilical hernia. (This does not include small umbilical hernias that are fat containing only; subjects with this specific type of hernia are allowed in the study, and this type of hernia could be managed and closed primarily with closure of the surgical site.)

  24. Large ventral hernia.

  25. Use of insulin.

  26. Anticoagulation or antiplatelet therapies.

  27. History of gastrointestinal cancer.

  28. Limited life expectancy.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose control | 6 and 12 months after the procedure
  Change in blood glucose control, as measured by the average of two HbA1c values at 6-months and 12-months post-procedure and at other time points, compared to the average of two HbA1c values 1-month pre-procedure.
Lack of serious adverse events (SAEs) | Through 1 year study completion
  Lack of serious adverse events (SAEs) assessed continuously during or after the procedure

SECONDARY OUTCOMES:
Change in Insulin Sensitivity | 6 and 12 months after the procedure
  Change in insulin sensitivity as measured by hyperinsulinemic euglycemic clamp at 6 and 12 months, as compared to pre-procedure
Change in blood glucose control | 1-week, 3, 6, and 12-months post procedure
  Change in blood glucose control (time in range, etc.) as measured by Continuous Glucose Monitoring (CGM) pre-procedure, and at 1-week, 3, 6 and 12-months post procedure
Change in fasting plasma glucose (FPG) | 1, 3, 6, and 12-month post procedure
  Change in fasting plasma glucose (FPG) and mean glycemic excursion as measured by oral glucose tolerance test (OGTT) pre-procedure and 1, 3, 6 and 12-months post procedure
Reduction in body weight | 1, 2, 3, 4, 10, 12, 18 weeks, and 6, 8, 10, 12 months post procedure
  Reduction in body weight measured at each clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas; Mark Andrew, MD, Study Director — Medality Medical
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The research team will send deidentified study results to Medality Medical

REFERENCES:
- [Background] Andrew MS, Huffman DM, Rodriguez-Ayala E, Williams NN, Peterson RM, Bastarrachea RA. Mesenteric visceral lipectomy using tissue liquefaction technology reverses insulin resistance and causes weight loss in baboons. Surg Obes Relat Dis. 2018 Jun;14(6):833-841. doi: 10.1016/j.soard.2018.03.004. Epub 2018 Mar 9. PMID 29631983